CLINICAL TRIAL: NCT01030120
Title: A 6 Week Randomized, Double Blind, Placebo-controlled Study With a 6 Week Open Label Extension to Assess the Efficacy of Etanercept in the Treatment of Chronic Idiopathic Urticaria
Brief Title: Etanercept for the Treatment of Chronic Urticaria
Acronym: EtanerceptCIU
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to complete agreement with sponsor
Sponsor: University of Utah (Other)
Responsible Party: Christopher Hull, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36414
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Idiopathic Urticaria
Keywords: chronic idiopathic urticaria; etanercept
MeSH Terms: conditions — Chronic Urticaria | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- etanercept (Active Comparator): etanercept 50mg BIW
  Interventions: Drug: etanercept
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: etanercept — etanercept 50mg BIW S.Q.
  Other Names: enbrel
  Arms: etanercept
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of etanercept for patients with chronic idiopathic urticaria unresponsive to antihistamines.

DETAILED DESCRIPTION:
Chronic urticaria is a common condition which can be debilitating, difficult to treat, and sometimes life-threatening. Approximately 15-25% of the population is affected by urticaria at least once in their lifetime, and chronic urticaria develops in more than 25% of these cases. Chronic urticaria is characterized by frequent, often daily, development of pruritic wheals of 6 weeks duration or longer. The average duration of chronic urticaria is 3-5 years in adults. In the majority of cases, an underlying trigger for the urticaria is not identified and these cases are referred to as idiopathic (CIU). These considerations have led to the hypothesis that CIU may have an autoimmune etiology.

CIU is a major affliction causing serious disability to a degree equal to that experienced by sufferers from coronary artery disease. Antihistamines are the most common therapy used. However, most cases of CIU are resistant to combinations of antihistamines and other therapies. In addition, patients are often intolerant to the side effects of antihistamines including sedation and cognitive dysfunction. The treatment of CIU patients can be frustrating. For those who do not respond to typical treatments, other therapies are needed. In many patients, immunosuppressant medications are required but this can lead to adverse effects such as renal dysfunction, liver function abnormalities, and anemia. A safer and more efficacious therapy is clearly needed for CIU.

A few preclinical investigations have demonstrated an upregulation of TNF-alpha in patients with CIU. This is in contrast to acute urticaria where TNF-alpha does not appear to play as important of a role in the inflammatory response . This may explain why patients with CIU do not typically respond to usual therapies for acute urticaria. It has been suggested that CIU is an immediate hypersensitivity phenomenon appearing immediately after exposure to an antigen, but the presence of a delayed inflammatory phase is nevertheless observed in this pathology. Soluble factors play a role in this delayed inflammatory phase. Cytokines, including TNF-alpha, are important mediators the pathogenesis of this delayed response. Studies have demonstrated a similar immune profile as that found in patients with rheumatoid arthritis. In one study, cytokines were evaluated in lesional and non-lesional skin of patients with acute urticaria, CIU, delayed pressure urticaria, and cold urticaria. This study demonstrated upregulation of TNF-alpha on endothelial cells and perivascular cells in the dermis. Additionally, TNF-alpha was expressed throughout the epidermis in lesional and non-lesional skin of CIU patients, but not controls. These preclinical investigations support the use of targeted therapy of TNF-alpha in patients with CIU. Therapies directed at modulating the effects of TNF-alpha, including etanercept, may provide effective and safe long-term treatment for patients not responding to anti-histamines alone.

HYPOTHESIS: We hypothesize that the blockage of TNF with etanercept could be a useful and safe therapy for patients with CIU.

OBJECTIVES:

Primary Objective: To determine the efficacy of etanercept on the clinical features of CIU. A positive response to treatment (a % change from baseline of urticaria activity scores

Secondary Objective: Study the safety of etanercept in the treatment of CIU

ELIGIBILITY:
Inclusion Criteria:

1. History of CIU occurring at least biweekly for greater than 6 week
2. Adult subjects between the ages of 18-70 years
3. Failure to respond to systemic antihistaminic therapy
4. Negative TB skin testing at baseline
5. Subjects willing to comply with study requirements
6. Negative urine pregnancy test at enrollment
7. Voluntarily sign and date informed consent form

Exclusion Criteria:

1. Current enrollment in any other investigational device or investigational drug trial(s), or receipt of any other investigational agent(s) within 28 days before baseline visit.
2. Known hypersensitivity to Enbrel® (etanercept) or any of its components or known to have antibodies to etanercept.
3. Latex sensitivity
4. Prior or concurrent use of cyclophosphamide therapy
5. Concurrent sulfasalazine therapy.
6. Known HIV-positive status or known history of any other immuno-suppressing disease.
7. Any mycobacterial disease or high risk factors for tuberculosis (TB), such as family member with TB, positive purified protein derivative (PPD) or taking anti-tuberculosis medication
8. Active or chronic infection within 4 weeks before screening visit, or between the screening and baseline visits.
9. Severe comorbidities (diabetes mellitus requiring insulin; CHF of any severity or myocardial infarction or cerebrovascular accident or transient ischemic attack within 3 months of screening visit; unstable angina pectoris, uncontrolled hypertension (sitting systolic BP <80 mm Hg or > 160 or diastolic BP > 100 mm Hg), oxygen-dependent severe pulmonary disease, history of cancer within 5 years [other than resected cutaneous basal or squamous cell carcinoma of the skin or in situ cervical cancer])
10. Exposure to hepatitis B or hepatitis C or to high risk factors for hepatitis B or C, such as intravenous drug use in patient.
11. Systemic lupus erythematosus, history of multiple sclerosis, transverse myelitis, optic neuritis or seizure disorder.
12. Use of a live vaccine 90 days prior to screening visit, or concurrent use of a live vaccine..
13. Any condition or circumstances judged by the patient's investigator to render this clinical trial detrimental or otherwise unsuitable for the patient's participation.
14. History of non-compliance with other therapies.
15. Concurrent use of anakinra.
16. Use of systemic immunosuppressive medication within 2 weeks of enrollment
17. Use of dapsone, sulfapyridine, sulfasalazine, or colchicine within 2 weeks of enrollment
18. Use of systemic corticosteroid within 2 weeks of enrollment
19. For females of childbearing potential, a refusal to use an acceptable form of contraceptive including oral or patch birth control, injectable birth control, intrauterine device, surgical sterilization, condom, barrier, or spermicide, post-menopausal, or complete abstinence from sexual activity.
20. For females, pregnancy, breast-feeding, or lactation
21. Active or recent (within the previous month) infection by staphylococcus aureus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of etanercept on the clinical features of CIU. A positive response to treatment (a % change from baseline of urticaria activity scores | 12 weeks

SECONDARY OUTCOMES:
Study the safety of etanercept in the treatment of CIU | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hull, MD, Principal Investigator — University of Utah Department of Dermatology
Locations (1):
- University of Utah Department of Dermatology, Salt Lake City, Utah, United States